CLINICAL TRIAL: NCT02446366
Title: Phase I Dose-Escalation Study of Hypofractionated SBRT for Adjuvant/Salvage Radiotherapy in Prostate Cancer
Brief Title: Hypofractionated Stereotactic Body Radiation Therapy for Patients With Prostate Cancer That Was Removed by Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-14-8; NCI-2015-00296 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-14-8 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-05-18 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stage II Prostate Adenocarcinoma; Stage IIB Prostate Cancer; Stage III Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (hypofractionated SBRT) (Experimental): Patients undergo 5, 10, or 15 fractions of hypofractionated SBRT daily over 1-3 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo hypofractionated SBRT
  Other Names: SBRT

SUMMARY:
This phase I trial studies the side effects and the best dose of hypofractionated stereotactic body radiation therapy (SBRT) in treating patients with prostate cancer that was removed by surgery. Hypofractionated SBRT delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and may have fewer side effects than standard radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine maximum tolerated dose-per-fraction for SBRT to the prostate fossa following prostatectomy based on acute toxicity (< 90 days).

SECONDARY OBJECTIVES:

I. To describe the acute (< 90 days) toxicities and adverse events associated with hypofractionated SBRT when administered to the prostate bed in the post-prostatectomy setting.

II. To describe the late (> 90 days from treatment) toxicities and adverse events associated with hypofractionated SBRT when administered to the prostate bed in the post-prostatectomy setting.

TERTIARY OBJECTIVES:

I. To describe the patient-reported toxicity/quality of life (QOL) following hypofractionated SBRT treatment.

OUTLINE: This is a dose-escalation study.

Patients undergo 5, 10, or 15 fractions of hypofractionated SBRT daily over 1-3 weeks.

After completion of study treatment, patients are followed up at 2, 6, and 13 weeks and then at 6, 9, 12, 18, 24, 30 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate treated primarily with radical prostatectomy

  * Any type of radical prostatectomy is permitted including retropubic, perineal, laparoscopic or robotically assisted; there is no time limit for the date of radical prostatectomy
* One of the following pathologic classifications

  * T3N0 disease with or without a positive surgical margin or
  * T2N0 disease with or without a positive surgical margin

    * Those with T2N0 disease and a negative margin must have a detectable prostate-specific antigen (PSA) following radical prostatectomy or
    * Must have had an undetectable PSA after prostatectomy and has since had a rise in post-operative PSA to 0.2 ng/mL or greater
* Zubrod performance status of 0 -1
* No distant metastases, based on the following workup within 60 days prior to registration

  * Magnetic resonance imaging (MRI) of the pelvis
  * Bone scan or sodium fluoride positron emission tomography (PET), that if suspicious has MRI or plain X-rays to rule out bone metastasis
* Patients can be on androgen deprivation therapy
* Ability to understand and willingness to sign a study-specific informed consent prior to study entry

Exclusion Criteria:

* N1 patients are ineligible, as are those with lymph node (LN) enlargement > 1.5 cm by computed tomography (CT) or MRI of the pelvis, unless the LN is biopsy proven to be negative
* Gross residual disease in the prostate fossa appreciated wither on digital rectal examination (DRE) or on imaging, unless biopsy proven not to contain cancer
* Patients who were exposed to neoadjuvant chemotherapy or chemotherapy after prostatectomy
* Prior radiation of any kind to the prostate gland or pelvis

  * Prior brachytherapy is not allowed
* History of inflammatory colitis or other active severe comorbidities
* Patients who are on immunosuppressant medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2023-02-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose-per-fraction based on acute toxicity assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.03 | < 90 days
  Maximum tolerated dose (MTD) is defined as the highest dose tested in which none or only one patient experienced dose limiting toxicity (DLT) attributable to the radiation therapy when 12 patients were treated at that dose and are evaluable for toxicity and is one dose level below the lowest dose level tested where two or more patients experienced radiation associated DLT. All toxicities and side effects of all patients who start SBRT will be recorded and summarized.

SECONDARY OUTCOMES:
Incidence of adverse events assessed according to CTCAE v. 4.03 | Up to 36 months after completion of SBRT
  All toxicities and side effects of all patients who start SBRT will be recorded and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ballas, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Ballas LK, Luo C, Chung E, Kishan AU, Shuryak I, Quinn DI, Dorff T, Jhimlee S, Chiu R, Abreu A, Jennelle R, Aron M, Groshen S. Phase 1 Trial of SBRT to the Prostate Fossa After Prostatectomy. Int J Radiat Oncol Biol Phys. 2019 May 1;104(1):50-60. doi: 10.1016/j.ijrobp.2018.12.047. Epub 2018 Dec 31. PMID 30605751